CLINICAL TRIAL: NCT02737527
Title: Comparison of the Efficacy of the Ultrasound With Fluoroscopy in Guidance of Lumbar Sympathetic Block: A Prospective Randomized Open-label Trial
Brief Title: Comparison of the Efficacy of the Ultrasound With Fluoroscopy in Guidance of Lumbar Sympathetic Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Clinical Associate Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1510-130-716
Record Dates: First submitted 2016-03-25; First posted 2016-04-14 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Complex Regional Pain Syndrome; Postherpetic Neuralgia; Diabetic Polyneuropathy; Peripheral Neuropathy
Keywords: ultrasound; lumbar sympathetic block
MeSH Terms: conditions — Complex Regional Pain Syndromes; Neuralgia, Postherpetic; Diabetic Neuropathies; Peripheral Nervous System Diseases | interventions — Ultrasonography; Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound with Fluoroscope (Experimental): This group undergoes lumbar sympathetic block using ultrasound and fluoroscope.
  Preparation: Inserts 24G intravenous route for Lumbar Sympathetic Block (LSB) Device: Uses 15-cm Chiba needle for Lumbar Sympathetic Block (LSB) Device: Uses Ultrasound for Lumbar Sympathetic Block (LSB) Drug: 10 ml of 0.25% levobupivacaine injection for LSB Intervention: Temperature measurement for Lumbar Sympathetic Block (LSB) Intervention: Postprocedure care for LSB
  Interventions: Procedure: 24G intravenous route for Lumbar Sympathetic Block (LSB):; Device: 15-cm Chiba needle for Lumbar Sympathetic Block (LSB); Device: Ultrasound for Lumbar Sympathetic Block (LSB); Drug: 10 ml of 0.25% levobupivacaine injection for LSB; Procedure: Temperature measurement for Lumbar Sympathetic Block (LSB); Procedure: Postprocedure care for LSB
- Fluoroscope only (Active Comparator): This group undergoes lumbar sympathetic block using fluoroscope only.
  Device: Inserts 24G intravenous route for Lumbar Sympathetic Block (LSB) Device: Uses 15-cm Chiba needle for Lumbar Sympathetic Block (LSB) Device: Uses Fluoroscope for Lumbar Sympathetic Block (LSB) Drug: 10 ml of 0.25% levobupivacaine injection for LSB Intervention: Temperature measurement for Lumbar Sympathetic Block (LSB) Intervention: Postprocedure care for LSB
  Interventions: Procedure: 24G intravenous route for Lumbar Sympathetic Block (LSB):; Device: 15-cm Chiba needle for Lumbar Sympathetic Block (LSB); Device: Fluoroscope for Lumbar Sympathetic Block (LSB); Drug: 10 ml of 0.25% levobupivacaine injection for LSB; Procedure: Temperature measurement for Lumbar Sympathetic Block (LSB); Procedure: Postprocedure care for LSB

INTERVENTIONS:
Procedure: 24G intravenous route for Lumbar Sympathetic Block (LSB): — Enrolled subjects enter the operative room with a 24G intravenous route, and then non-invasive blood pressure and pulse oxygen saturation level are continuously monitored during and after the procedure.
  Other Names: lumbar sympathetic ganglion block (LSGB); lumbar sympathetic chain block
Device: 15-cm Chiba needle for Lumbar Sympathetic Block (LSB) — The skin entry point is infiltrated using 1% lidocaine. A curved 21 G, 15-cm Chiba needle (Cook Inc., Bloomington, IN, USA) is then advanced toward the anterolateral edge of target vertebral body by posterolateral approach in patients with prone position.
Device: Ultrasound for Lumbar Sympathetic Block (LSB) — Using Ultrasound, the L3 is identified by locating the lumbosacral junction on a paramedian sagittal scan and then counting cranially. After marking the level of L3 vertebra, the modified transverse scan through lumbar intertransverse space (ITS) is obtained with the transducer positioned 4-6 cm lateral to the mid-line at the L2-L3 intervertebral level. The needle is inserted from a lateral to medial direction using in-plane technique. The needle tip is inserted towards the anterior fascia of the psoas major muscle as close as paravertebral space.
  Arms: Ultrasound with Fluoroscope
Device: Fluoroscope for Lumbar Sympathetic Block (LSB) — Briefly, fluoroscopic guided LSBs are performed at the lower third of the L2 or the upper third of the L3 vertebra. A targeted lumbar vertebral is identified by AP fluoroscopic imaging and the fluoroscopic C-arm is adjusted 25-35° laterally to avoid the transverse process over the needle pathway. After the skin infiltration, the needle is advanced toward the anterolateral edge of the target lumbar vertebra under fluoroscopic guidance using the tunnel vision technique.
  Arms: Fluoroscope only
Drug: 10 ml of 0.25% levobupivacaine injection for LSB — After excluding vascular injection with contrast media by a C-arm image intensifier on anteroposterior (AP) and lateral view, 10 ml of 0.25% levobupivacaine is injected through the Chiba needle.
Procedure: Temperature measurement for Lumbar Sympathetic Block (LSB) — Temperature monitoring and measurement: skin-surface temperatures are monitored with small, adhesive thermocouple probes attached bilaterally to the plantar surface of the feet using transparent patches at 1-min intervals for a maximum of 20 min.
Procedure: Postprocedure care for LSB — Adverse events such as genitofemoral nerve block, lumbar plexus block (transient unilateral leg weakness), or others are documented during and after the procedure for 30 min.

SUMMARY:
This study compares the efficacy of the ultrasound with fluoroscope in guidance of lumbar sympathetic block (LSB). The goals of the study are; 1) To show that US-guided LSB results in shorter performance time compared to fluoroscope-guided LSB, 2) To evaluate the efficacy and safety of US-guided LSB, and 3) To verify that US-guided LSB has similar success rates to fluoroscope-guided LSB. 50 patients who are supposed to undergo LSB due to sympathetically maintained pain, satisfy criteria of inclusion and exclusion, and voluntarily sign the informed consent will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have sympathetically-mediated pain and are supposed to undergo LSB procedure (e.g. pain with asymmetric skin temperature of lower limb in previous thermography, small fiber disorder in previous quantitative sudomotor axon reflex test (QSART), vascular insufficiency in lower extremities, diabetic polyneuropathy, postherpetic neuralgia, complex regional pain syndrome, cancer-related neuropathic pain such as chemotherapy-induced peripheral neuropathy, other lower extremity neuropathies, lower extremity crush injury etc.)
* Numeric rating scale (NRS) ≥ 4/10
* Failure of previous conservative treatments, such as physiotherapy, oral medication, or other noninvasive treatment

Exclusion Criteria:

* Previous lumbar sympathetic neurolysis
* Bleeding tendency
* Local infection
* Allergy to local anesthetics or contrast media
* Pregnancy
* Severe variation near procedure site-scoliosis, tumor, abdominal aneurysm, etc.
* BMI ≥ 30 kg/m2
* Cognitive dysfunction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Difference in Procedure time (I1) | through the LSB procedure completion (day 0)
  U group: the time interval between the contact of the US probe with the patient's skin and the completion of the injection of levobupivacaine F group: the time interval between the first radiographic image and the end of the injection of levobupivacaine

SECONDARY OUTCOMES:
Success rate | through the LSB procedure completion (day 0)
  Definition of successful LSB: temperature rises as high as 2℃ from initial temperature on an ipsilateral sole in 20 min after the injection of levobupivacaine.
  Temperatures are measured at 1-min intervals and recorded from the time of administration of levobupivacaine onwards. Assessments are continued for a maximum of 20 min.
Onset time of block (I2) | through the LSB procedure completion (day 0)
  Definition of successful LSB: temperature rises as high as 2℃ from initial temperature on an ipsilateral sole in 20 min after the injection of levobupivacaine.
  Temperatures are measured at 1-min intervals and recorded from the time of administration of levobupivacaine onwards. Assessments are continued for a maximum of 20 min.
The number of needle passes | through the LSB procedure completion (day 0)
  In both groups, the initial needle insertion counted as one pass; any subsequent needle advancement that is preceded by a withdrawal of more than 1 cm counts as an additional pass
The number of the needle contact to bone during the procedure | through the LSB procedure completion (day 0)
Spreading pattern of contrast dye during the procedure | through the LSB procedure completion (day 0)
  Spreading pattern of contrast dye will be measured by 3 patterns (normal/muscular spread pattern/ intravascular spreading).
An 11-pointed NRS pain score related to the procedure only | through the LSB procedure completion (day 0)
  measured twice -1) just after the procedure at OR, and 2) at recovery room just before discharge
Any adverse events | Up to 72 hours after the procedure
  genitofemoral nerve block, lumbar plexus block (transient unilateral leg weakness, or other events
Changes of an 11-pointed NRS pain score from baseline for their lower extremity pain | performs telephone follow-up in 72 hours.
Procedure-related NRS pain score | performs telephone follow-up in 72 hours.
Changes of dose in analgesics | performs telephone follow-up in 72 hours.
  NSAIDs, paracetamol, and opioids
Any adverse events remained | performs telephone follow-up in 72 hours.
A 5-pointed Likert satisfaction scale related to the procedure | performs telephone follow-up in 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Ryu JH, Lee CS, Kim YC, Lee SC, Shankar H, Moon JY. Ultrasound-Assisted Versus Fluoroscopic-Guided Lumbar Sympathetic Ganglion Block: A Prospective and Randomized Study. Anesth Analg. 2018 Apr;126(4):1362-1368. doi: 10.1213/ANE.0000000000002640. PMID 29189275